CLINICAL TRIAL: NCT05914636
Title: Evaluation of Intestinal Microbiota Implication in Ruptured Intracranial Aneurysm: a Comparison of Ruptured and Unruptured Patient With Taxonomic and Metabolic Evaluation of Microbiota
Brief Title: Evaluation of Intestinal Microbiota Implication in Ruptured Intracranial Aneurysm
Acronym: AneBiote
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0263; 2021-A02202-39 (Other: ID-RCB)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Intracranial Sacciform Aneurysm
Keywords: Intracranial aneurysm; intestinal microbiota; risk factor; ruptured
MeSH Terms: conditions — Intracranial Aneurysm; Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ruptured: Patient with a ruptured intracranial sacciform aneurysm for all location. The diagnosis of ruptured aneurysm is made on MRI, Angio-CT or digital substraction angiography with no doubt
  Interventions: Biological: analysis of foecal microbiota
- unruptured: Patient with an unruptured intracranial sacciform aneurysm for all location. The diagnosis of unuptured aneurysm is made on MRI, Angio-CT or digital substraction angiography with no doubt
  Interventions: Biological: analysis of foecal microbiota

INTERVENTIONS:
Biological: analysis of foecal microbiota — An analysis of foecal microbiota including taxonomic and metabolomic analysis will be performed and compared between ruptured and unruptured patient.
  confundens factors as diet, obesity for microbiota and as smoking, hypertension, size for aneurysm ruptured will be sampled and independence will be analyzed.

SUMMARY:
The physiopathology of intracranial aneurysm from initiation to ruptured is incompletely understood but included inflammation. The microbiota is known to interact with brain and can promote inflammation. The objective of this study is to describe microbiota with taxonomic and metabolomic analysis. A comparison between ruptured and unruptured intracranial aneurysm will be performed. The study hypothesis is that microbiota is different between ruptured and unruptured patient.

ELIGIBILITY:
Inclusion Criteria:

* one or more intracranial sacciform aneurysm ruptured or not in function of the inclusion group

Exclusion Criteria:

* Transient modification of microbiota: Antibiotherapy in the last 3 months, pre or probiotic in the last month, gastrostomy, ileostomy, bariatric surgery, digestive tract resection, gastro-duodenal ulcer surgery or during the last month, chronic inflammatory disease of the digestive tract (like Crohn), BMI for more than 30, Very restrictive diet (like vegan
* Specific pathologies increasing the incidence of aneurysm ( kidney autosomic dominant polycystosis, Type 1 neurofibromatosis, Rendu-Osler, MArfan
* Participation to a study with the objective of microbiota modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with ruptured aneurysm and unruptured aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Taxonomic faecal microbiota description | The faecal samples will be taken at 3 days+/-2 after the ruptured and during the arteriography for the unruptured group within 3 months after inclusion
  The results of the taxonomic analysis of fecal samples will be described in the two groups. Interesting parameter will be selected for further analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dumot Chloé, Dr PhD, Principal Investigator — Hôpital neurologique P. Wertheimer